CLINICAL TRIAL: NCT04272710
Title: Prognostic Characteristics Difference Between the Hypertension Patients With and Without ACEI Treatment When Suffered With 2019-nCoV Infection in China
Brief Title: Prognositc Factors in COVID-19 Patients Complicated With Hypertension
Status: Withdrawn | Type: Observational
Why Stopped: Similar projects have been registered, and it need to be withdrawn.
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Associate Professor, Chongqing Medical University
Other Study IDs: 2020-02
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACEI treatment: hypertension patients with ACEI treatment when suffered with novel coronavirus infection in China
- Control: hypertension patients without ACEI treatment when suffered with novel coronavirus infection in China

SUMMARY:
There are currently no clinical studies reporting clinical characteristics difference between the hypertension patients with and without ACEI treatment when suffered with novel coronavirus infection in China.

DETAILED DESCRIPTION:
At present, the outbreak of the new coronavirus (2019-nCoV) infection in Wuhan and Hubei provinces has attracted great attention from the medical community across the country. Both 2019-nCoV and SARS viruses are coronaviruses, and they have a large homology.

Published laboratory studies have suggested that SARS virus infection and its lung injury are related to angiotensin-converting enzyme 2 (ACE2) in lung tissue. And ACE and ACE2 in the renin-angiotensin system (RAS) are vital central links to maintain hemodynamic stability and normal heart and kidney function in vivo.

A large amount of evidence-based medical evidence shows that ACE inhibitors are the basic therapeutic drugs for maintaining hypertension, reducing the risk of cardiovascular, cerebrovascular, and renal adverse events, improving quality of life, and prolonging life in patients with hypertension. Recent experimental studies suggest that treatment with ACE inhibitors can significantly reduce pulmonary inflammation and cytokine release caused by coronavirus infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old;
* Diagnosed with 2019-nCoV. Diagnostic criteria including: Laboratory (RT-PCR) confirmed 2019-nCoV infection; CT of the lung conformed to the manifestation of viral pneumonia.
* Diagnosed with primary hypertension.
* Criteria for severe or critical ill conditions: Respiratory rate >=30/min; or Rest SPO2<=93%; or PaO2/FiO2<=300mmHg.

Exclusion Criteria:

* Near-death state (expected survival time less than 24 hours);
* Malignant tumor;
* Pregnancy or puerperium women;
* ACEI contraindication
* Patients who refused to participant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the hypertension patients with and without ACEI treatment when suffered with novel coronavirus infection in China
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Occupancy rate in the intensive care unit (ICU) | up to 28 days
  The percentage of patients admitted to the ICU at any time during the 28 days of onset COVID-19.
Mechanical Ventilation | up to 28 days
  The number of patients requiring mechanical ventilation.
Death | up to 28 days
  The number of patients who died of 2019-nCoV infection.

SECONDARY OUTCOMES:
All cause mortality | up to 28 days
  The number of died 2019-nCoV infected patients from any cause.
Time from onset of symptoms to main outcome and its components | up to 28 days
  Time from onset of symptoms to admitted to the ICU, requiring mechanical ventilation, and death.
Time to Clinical Recovery | up to 28 days
  Time to Clinical Recovery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China